CLINICAL TRIAL: NCT01800617
Title: Phase II Single Daily-Dose Response Study of a New Liothyronine Sodium (T3) Preparation With Sustained Effects in Hypothyroid Patients
Brief Title: A Study of T3 Therapy in Patients With Hypothyroidism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipe, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCT303-2
Record Dates: First submitted 2013-02-18; First posted 2013-02-27 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liothyronine, Sodium (Experimental)
  Interventions: Drug: Liothyronine, Sodium

INTERVENTIONS:
Drug: Liothyronine, Sodium

SUMMARY:
The purpose of this study is to test a new thyroid hormone preparation. The thyroid gland produces two thyroid hormones: mostly T4 and a smaller amount of T3. Thyroid hormone therapy for hypothyroidism or thyroid cancer is generally provided using levothyroxine, which is a synthetic form of T4. T4 is converted into the active hormone T3 in the circulation. Therefore, some researchers believe that T3 levels in T4-treated patients may be slightly lower than in individuals whose own thyroid gland is functioning normally. Symptoms of hypothyroidism have been suggested to occur because of this possible T3 deficiency, although this is controversial. Studies of T3, added to or substituted for T4 in traditional levothyroxine regimens, have generally not shown any benefit of T3. However, it is still possible that no benefit is seen because of the short duration of action or "half-life" of T3. This short-life makes it necessary to dose T3 twice or three times daily. Despite multiple daily doses of T3, T3 levels during its therapy tend to be troubled by peaks and troughs. These peaks can be associated with symptoms of excessive thyroid hormone levels. This study will look at TSH and thyroid hormone levels following a daily dose of a new preparation of T3 that may have longer duration of action than liothyronine. This preparation of T3 is called Thyromax® or BCT303. The investigators believe that steady levels of T3 will be seen after taking Thyromax®. The investigators believe that in patients with hypothyroidism use of Thyromax® in the correct dose will produce normal TSH levels, without producing symptoms of too much thyroid hormone. The goal of future studies is to test whether Thyromax® may be a potential treatment for hypothyroidism, by comparing it with traditional levothyroxine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Hypothyroid patients taking levothyroxine
* Age 18-65
* Able to make weekly in-person visits to Washington, D.C.

Exclusion Criteria:

* Pregnancy or lactation
* Chronic medical conditions such as heart disease or any other chronic medical conditions such as lung disease (e.g. asthma), kidney disease (e.g. kidney failure), liver disease (e.g. hepatitis), diabetes, or cancer.
* Steroid medications such as estrogen, progesterone, estrogen or progesterone related medications, testosterone, or glucocorticoids
* Already taking T3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Measurement of Blood Levels of Thyroid Hormone Sensitive Parameters | Six Weeks.
  Serum Total T3, TSH

SECONDARY OUTCOMES:
Measurement of Oxygen Consumption | Six Weeks.
  Resting Metabolic Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States